CLINICAL TRIAL: NCT00003502
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Stage II, III, or IV Mantle Cell Lymphoma
Brief Title: Antineoplaston Therapy in Treating Patients With Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-LY-9; CDR0000066542 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Contiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Mantle Cell Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — antineoplaston A10; antineoplaston AS 2-1; Biological Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: antineoplaston AS2-1
Procedure: alternative product therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: complementary and alternative therapy
Procedure: differentiation therapy

SUMMARY:
RATIONALE: Antineoplastons are naturally-occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial is studying how well antineoplaston therapy works in treating patients with stage II, stage III, or stage IV mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and possible effectiveness of antineoplastons A10 and AS2-1 in patients with serious or immediately life-threatening stage II, III, or IV mantle cell lymphoma.
* Evaluate the response to, tolerance to, and side effects of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive gradually escalating doses of antineoplaston A10 and antineoplaston AS2-1 intravenously 6 times daily until the maximum tolerated dose is reached. Treatment continues in the absence of disease progression or unacceptable toxicity.

Tumors are measured every 8 weeks for 6 months, every 3 months for 2 years, every 6 months for the third and fourth years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage II, III, or IV mantle cell lymphoma that is not curable by surgery, radiotherapy, and/or chemotherapy
* Measurable tumor of greater than 2 cm in largest diameter for lymph nodes located in head, neck, axillary, inguinal, and femoral areas (at least 1 cm for other areas)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC greater than 2000/mm^3
* Platelet count greater than 20,000/mm^3

Hepatic:

* No hepatic insufficiency
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No hypertension
* No history of congestive heart failure
* No history of cardiovascular conditions that contraindicate high dosages of sodium

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections requiring treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulatory agent (e.g., interferon or interleukin-2)

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agent

Endocrine therapy:

* At least 4 weeks since prior corticosteroids (e.g., dexamethasone or prednisone)
* No concurrent dexamethasone, prednisone, or other corticosteroids

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy
* No concurrent antibiotics, antifungals, or antivirals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States